CLINICAL TRIAL: NCT04796220
Title: Focused Ultrasound With Low-Dose Gemcitabine to Augment Immune Control of Early Stage Breast Cancer
Brief Title: Focused Ultrasound and Gemcitabine in Breast Cancer
Acronym: Breast 54
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Patrick Dillon, MD (Other)
Responsible Party: Sponsor-Investigator, Patrick Dillon, MD, Associate Professor, Department of Medicine, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200277
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm B: FUS (Experimental)
  Interventions: Device: Focused Ultrasound
- Arm C: GEM/FUS (Experimental)
  Interventions: Other: Gemcitabine and Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — Focused ultrasound will be applied to up to 2 breast lesions on day 8.
  Other Names: EchoPulse
  Arms: Arm B: FUS
Other: Gemcitabine and Focused Ultrasound — Gemcitabine (900 mg/m2) will be administered intravenously on day 1.Focused ultrasound will be applied to up to 2 breast lesions on day 8.
  Other Names: Gemzar, EchoPulse
  Arms: Arm C: GEM/FUS

SUMMARY:
This study will test the use of focused ultrasound ablation, low-dose gemcitabine (a chemotherapy) and the combination of focused ultrasound ablation plus low-dose gemcitabine in patients with early-stage breast cancers. We will be testing the effects of each of these regimens on cells in the immune system. We hypothesize that the combination of focused ultrasound ablation and gemcitabine will decrease myeloid-derived suppressor cells and will increase T cell activity. We also hypothesize that focused ultrasound ablation and low-dose gemcitabine will be safe and will result in non-inferior surgical completion rates and tumor margin assessments.

ELIGIBILITY:
Inclusion Criteria:

* Disease Status

  * Patients must have histologically confirmed, newly diagnosed breast cancer, stage 1-3 disease and be appropriate surgical candidates for complete resection. Recurrent disease patients must have disease localized to the breast, chest wall or axilla and must be surgical candidates for completion resection of recurrent disease.
  * If genomic profiling is performed, then the results must indicate that the cancer is high-risk
  * Any receptor status may be eligible (estrogen receptor, progesterone receptor, HER2 receptor)
  * Patients must have a lesion in the breast/chest wall/axilla that is accessible to focused ultrasound ablation.

Accessible is defined as the following:

* A targetable portion of the tumor must be ≥ 5mm from the skin
* The rib cage should not be in the prefocal ultrasound path or behind the target area of the lesion (minimum distance from the posterior aspect of the target area to rib cage must be at least 10 mm).

Participants must have at least one high-risk feature of breast cancer (tumor size and nodal status may be measured by mammogram, MRI, US, CT, or calipers):

* Triple negative breast cancer with Tumor size ≥10mm
* Lymph node involvement by imaging or biopsy (any receptor status, any size)
* Tumor size ≥ 20mm (estrogen receptor positive, HER2 negative)
* Tumor size ≥ 10mm (HER2 receptor positive, any ER status)
* Tumor size ≥ 10mm and Oncotype or Mammaprint high status (estrogen receptor positive, HER2 negative) *If patient has more than one tumor, then the treated tumor must have a high-risk feature (if 2 tumors meet high risk criteria), they may both be treated).

  * Willing and able to provide written consent
  * Stated willingness to comply with all study procedures and availability for the duration of the study.
  * Male or female, ≥ 18 years
  * Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
  * ECOG performance status of 0-2
  * Adequate organ function
  * Agreement to adhere to lifestyle considerations throughout the study duration

Exclusion Criteria:

* Received other treatment (standard or investigational) for their current breast cancer.
* Pregnant or lactating
* Diagnosis of immunodeficiency or receiving systemic steroid therapy within 7 days prior to enrollment with the following exceptions:

  * In patients with adrenal or pituitary insufficiency replacement steroid doses are allowed; however, daily doses of 10 mg or more of prednisone (or equivalent) per day administered parenterally or orally are not allowed in patients with normal adrenal and pituitary function.
  * Inhaled steroids (e.g.: Advair®, Flovent®, Azmacort®) are permitted at low doses (less than 500 mcg fluticasone per day, or equivalent).
  * Topical, nasal, and intra-articular corticosteroids are acceptable.
* Known allergic reactions to gemcitabine
* Breast implant on the side of the body that will receive HIFU application
* Known history of HIV (Patients with HIV will be excluded because immunotherapy may impact the T cell profiling as part of the biologic correlates and the natural history of the disease)
* Known active Hepatitis B virus or Hepatitis C virus
* Other malignancy other than basal cell carcinoma of the skin or squamous cell carcinoma of the skin that is undergoing potentially curative therapy, ductal carcinoma in situ (DCIS), or in situ cervical cancer
* Active infection requiring other systemic therapy
* Participants in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator.
* Any condition(s) or diagnosis, both physical or psychological, or physical exam finding that precludes participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with any ≥ grade 3 adverse event | Adverse events collected through 30 days after the last study treatment
  Adverse events as measured by CTCAE v5.0
Rate of participants experiencing a delay in surgery | Through month 7 (Follow-up visit 2)
  Rate of participants experiencing a delay in surgery, beyond day 26
Rate of positive margins following surgery | Day 22
  Number of participants who have positive tumor margins at the time of surgery

SECONDARY OUTCOMES:
The effect of the treatments on myeloid-derived suppressor cells (MDSC) and CD8+ T cells in the tumor microenvironment | Day 22
  MDSC/CD8 ratio in the tumor
The effect of the treatments on circulating activated T cells | Measured through 30 days after the last active treatment visit
  Proportion of activated T cells in the blood
The effects of the treatments on dendritic cells in the tumor microenvironment | Day 22
  Dendritic cell maturation in the tumor; we will stain cells using panels of markers for maturation and use multi-spectral immunohistochemistry and/or flow cytometry to characterize the dendritic cell populations.
Patient satisfaction with treatment regimen and surgery | through month 7
  Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) will be used to assess patient satisfaction with the treatment regimen and surgery; graded on a scale from 0 to 4 and scoring outcomes vary depending on the question that is being asked.
Patient and physician reported results on cosmesis | through month 7
  Harvard /NSABP/RTOG Breast Cosmesis Grading Scale will be used to assess cosmesis; graded is on a scale of 1 to 4 with a higher score indicating a poorer outcome.
Residual cancer burden | Day 22
  MD Anderson Residual Cancer Burden Calculator

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dillon, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No